CLINICAL TRIAL: NCT02108743
Title: Albuterol and Dynamic Hyperinflation in Idiopathic Pulmonary Arterial Hypertension
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: American Medical Association Foundation (Other)
Responsible Party: Principal Investigator, Matthew Lammi, Assistant Professor of Medicine, Section of Pulmonary and Critical Care, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB8603
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension.
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albuterol (Active Comparator): 2.5 mg of albuterol inhaled via jet nebulizer 15 minutes prior to symptom-limited maximal CPET.
  Interventions: Drug: Albuterol.
- Placebo (Placebo Comparator): Normal saline placebo inhaled via jet nebulizer 15 minutes prior to symptom-limited maximal CPET.
  Interventions: Drug: Normal saline placebo

INTERVENTIONS:
Drug: Albuterol. — 2.5 mg of albuterol inhaled via jet nebulizer 15 minutes prior to symptom-limited maximal CPET.
  Arms: Albuterol
Drug: Normal saline placebo — Placebo inhaled via jet nebulizer 15 minutes prior to symptom-limited maximal CPET.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if dynamic hyperinflation seen in patients with idiopathic pulmonary artery hypertension (iPAH) improves with albuterol therapy.

DETAILED DESCRIPTION:
Only a few small studies have evaluated the relationship between iPAH, expiratory flow limitation, and exercise dyspnea. While not all patients with iPAH demonstrate airway involvement, those who demonstrate dynamic hyperinflation (DH), defined as a variable and temporary increase in end-expiratory lung volume, report increased dyspnea with exertion on maximal testing. There is a continued need for adjuvant therapy in iPAH, and bronchodilators have the potential to ameliorate dyspnea during exercise, which could lead to improved quality of life in this disabling condition. This study will investigate the presence of airway involvement in this population as measured by dynamic hyperinflation, and if there is any improvement in function with the use of inhaled albuterol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater.
* Idiopathic Pulmonary Arterial Hypertension, or Familial Pulmonary Arterial Hypertension.
* Forced expiratory flow 75% (FEF75%) of ≤ 65% of predicted.

Exclusion Criteria:

* Clinical instability or change in medication therapy in preceding 3 months.
* Allergy or intolerance to inhaled albuterol.
* Body mass index > 30
* Active tobacco use, or > 10 pack-year smoking history.
* Lung disease other than pulmonary hypertension
* Forced expiratory volume in 1 second (FEV1) ≤ 80% of predicted.
* Pregnancy
* Inability to perform pulmonary function testing.
* Inability to perform cardiopulmonary exercise testing.
* Supplemental oxygen requirement.
* Inability to read and understand English.
* Historical 6-minute walk distance <150 meters

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
End-expiratory lung volume:total lung capacity (EELV/TLC) ratio at matched metabolic isowork. | up to 3 days
  Determined by measuring inspiratory capacity every 2 minutes during cardiopulmonary exercise test (CPET)

SECONDARY OUTCOMES:
Change in peak oxygen consumption with albuterol | Study days 2 and 3
  Measured at the end of CPET
Change in O2 pulse with albuterol. | Study days 2 and 3
  Measured throughout CPET and compared at matched metabolic isotimes
Exercise time | Study days 2 and 3
  Total ramped exercise time
Borg dyspnea score | Days 2 and 3
  Measured every 2 minutes throughout CPET

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Lammi, MD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- LSUHSC Interim Louisiana Hospital, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Meyer FJ, Ewert R, Hoeper MM, Olschewski H, Behr J, Winkler J, Wilkens H, Breuer C, Kubler W, Borst MM; German PPH Study Group. Peripheral airway obstruction in primary pulmonary hypertension. Thorax. 2002 Jun;57(6):473-6. doi: 10.1136/thorax.57.6.473. PMID 12037220
- [Background] Fernandez-Bonetti P, Lupi-Herrera E, Martinez-Guerra ML, Barrios R, Seoane M, Sandoval J. Peripheral airways obstruction in idiopathic pulmonary artery hypertension (primary). Chest. 1983 May;83(5):732-8. doi: 10.1378/chest.83.5.732. PMID 6839814
- [Background] Laveneziana P, Garcia G, Joureau B, Nicolas-Jilwan F, Brahimi T, Laviolette L, Sitbon O, Simonneau G, Humbert M, Similowski T. Dynamic respiratory mechanics and exertional dyspnoea in pulmonary arterial hypertension. Eur Respir J. 2013 Mar;41(3):578-87. doi: 10.1183/09031936.00223611. Epub 2012 Jul 12. PMID 22790921
- [Background] Spiekerkoetter E, Fabel H, Hoeper MM. Effects of inhaled salbutamol in primary pulmonary hypertension. Eur Respir J. 2002 Sep;20(3):524-8. doi: 10.1183/09031936.02.02572001. PMID 12358324